CLINICAL TRIAL: NCT01514721
Title: Assessing the Efficacy and Tolerability of Changing to DuoTrav® (Travoprost 0.004%/Timolol 0.5% BAK-Free Fixed Combination), as Replacement Therapy in Patients Previously on Prior Prostaglandin Fixed Combination
Brief Title: Efficacy of Changing to DuoTrav® (Travoprost 0.004%/Timolol 0.5% BAK-Free Fixed Combination) From Prior Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-11-171
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma
Keywords: Open-angle glaucoma; Ocular hypertension; Pigment dispersion glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DuoTrav (Experimental): Travoprost/Timolol Maleate BAK-Free Fixed Combination, 1 drop self-administered in treated eye(s) once a day for 12 weeks
  Interventions: Drug: Travoprost/Timolol Maleate BAK-Free Fixed Combination

INTERVENTIONS:
Drug: Travoprost/Timolol Maleate BAK-Free Fixed Combination — Commercially marketed Travoprost/Timolol BAK-free ophthalmic solution indicated for the treatment of patients with open angle glaucoma (OAG) or ocular hypertension (OH).
  Other Names: DuoTrav®

SUMMARY:
The purpose of this study is to assess efficacy and tolerability of changing to DuoTrav® (Travoprost 0.004%/Timolol 0.5% BAK-free) from prior Xalacom® or Ganfort® fixed combination pharmacotherapy in patients with open-angle glaucoma or ocular hypertension with uncontrolled intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, open-angle glaucoma, or pigment dispersion glaucoma in both eyes.
* On a stable IOP-lowering regimen of prostaglandin fixed combination (either Xalacom or Ganfort) within 4 weeks prior to the Screening Visit.
* IOP between 19 and 35 mmHg at any time of day in at least 1 eye.
* Best corrected visual acuity (BCVA) of 6/60 (20/200 Snellen; 1.0 LogMAR) or better in each eye.
* Willing to discontinue the use of all other ocular hypotensive medication(s) prior to receiving the study medication for the entire course of the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity, or poor tolerance to any component of DuoTrav® deemed clinically significant in the opinion of the Principal Investigator.
* Corneal dystrophies in either eye.
* Risk of visual field or VA worsening as a consequence of participation in the study, in the investigator's best judgment.
* Any disease or condition that would preclude the safe administration of a topical beta-blocker, present a special risk to the subject, or interfere with optimal participation in the study.
* Women who are pregnant or lactating.
* Participation in any other investigational study within 30 days prior to the Screening Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in intra-ocular pressure (IOP) at final visit from prior therapy (i.e., from baseline) | 12 weeks
  Goldmann applanation tonometry will be performed at the baseline visit and the 12-week visit to record IOP. Change in IOP will be calculated. IOP will be measured in mmHg.

SECONDARY OUTCOMES:
Percentage of patients who reach target IOP (≤18mmHg) | 12 weeks
  Goldmann applanation tonometry will be performed at the 12-week visit to record IOP. Percentage of patients who reach target IOP will be calculated by comparing patients with IOP ≤18mmHg to the overall study population.
Change in Ocular Surface Disease Index (OSDI) score at final visit from baseline | 12 weeks
  An OSDI questionnaire will be completed by the subject at the baseline visit and at the 12-week visit. For each visit, an overall OSDI score will be calculated using individual item responses, and the change in OSDI score from baseline will be calculated.
Change in ocular hyperemia score at final visit from baseline | 12 weeks
  Ocular hyperemia will be assessed by qualified personnel at the baseline visit and again at the 12-week visit, and change from baseline will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Abayomi Ogundele, PharmD, Study Director — Alcon Research
Locations (1):
- Alcon Investigational Site, São Paulo, Brazil